CLINICAL TRIAL: NCT03763734
Title: High-Dose Steroids in High Pain Responders Undergoing Total Knee-arthroplasty: A Randomized Double Blinded Controlled Trial
Brief Title: High-Dose Steroid for Knee Arthroplasty Patients Expected to Have Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Niklas Ingemann Nielsen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBF_HK_02_2018
Record Dates: First submitted 2018-11-28; First posted 2018-12-04 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Knee Osteoarthritis; Perioperative/Postoperative Complications; Surgery; Opioid Use; Catastrophizing Pain; Chronic Pain
Keywords: Knee Arthroplasty; Knee Replacement; Perioperative Medicine
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Osteoarthritis, Knee; Postoperative Complications; Chronic Pain | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: A randomized double blinded controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All intervention drugs will be blinded by a nurse who is not a participant in the study or in the treatment of the patient in any way.
  The Patient, the administrator of the drug(nurse or doctor), the assessor, the investigator and the care team will all be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose Dexamethasone (Experimental): An intravenous bolus dose of Dexamethasone 1 mg/kg bodyweight administered preoperatively before surgery.
  Interventions: Drug: Dexamethasone
- Medium dose Dexamethasone (Active Comparator): An intravenous bolus dose of Dexamethasone 0,3 mg/kg bodyweight administered preoperatively before surgery.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — An intravenous bolus dose of dexamethasone given prior to surgery.
  Other Names: Dexa-ratiopharm

SUMMARY:
The purpose of the Study is to test a higher dose of steroids(Dexamethasone) given just prior to surgery in the setting of Fast-Track Knee surgery with Arthroplasty in a group of expected High Pain Responders and the effect on postoperative pain and postoperative inflammation.

DETAILED DESCRIPTION:
This study compares a new High-Dose dosage of steroids in the treatment of postoperative pain after Knee Arthroplasty in a Fast-Track setting in a group of expected High Pain Responders.

The investigators compare the already used dose(medium dose) with a new high dose(HD) steroid given as an intravenous bolus after the spinal anaesthesia has been given, but before the surgery starts.

The hypothesis is that by attenuating the inflammatory response to the surgery itself by the steroid Dexamethasone, the investigators expect a reduction in postoperative pain upon ambulation 24 hours after unilateral Knee Arthroplasty.

Patients referred to Unilateral Total KneeArthroplasty because of knee-osteoarthritis at Hvidovre Hospital, Capital Region of Denmark or Vejle Hospital, South Region of Denmark are screened and offered inclusion in the study.

The two groups will be randomized and double blinded. One group will be treated, as the current guideline in the investigator's Orthopedic fast-track Arthroplasty center, with the medium dose of steroid (0,3 mg dexamethasone/kg bodyweight).

The other group wil be treated with a high dose of steroid (1,0 mg dexamethasone/kg bodyweight).

The patients will be monitored the first 7 days after surgery, during the admission to the hospital, and by a Pain-diary in the patients own home.

Blood tests will be taken preoperatively and postoperatively to determine the effect of the highdose steroid on the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 90.
* Booked for unilateral knee-arthroplasty.
* Is able to take part in the investigation(selfreported pain and nausea/vomiting)
* Understands Danish or English, or has a translator available.
* Signed written consent.
* A daily use of 30 mg or more of morphine or morphine equivalents .
* A pain catastrophizing scale(PCS) score of >20.

Exclusion Criteria:

* Insulin-dependent diabetes melitus.
* Ongoing treatment with systemic glucocorticoids or immunosuppressing treatment(apart from inhaled glucocorticoids).
* Pregnancy/Breastfeeding
* Allergies for the investigational drug.
* A history of schizophrenia or bipolar diseases, or patients with permanent use of antipsychotic medication.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after 24 hours: VAS | 24 hours
  The amount of patients with moderate postoperative pain in a 5 meter walk test 24 hours postoperatively after total knee-arthroplasty.
  Pain is monitored by the Visual Analog Scale(VAS) 0-100 mm, where 0 is no pain and 100 mm is the worst pain. Moderate pain is considered a VAS >30 mm.

SECONDARY OUTCOMES:
Postoperative opioid usage | 7 days
  The amount of rescue opioids given in the postoperative period, and until 7 days after surgery.
Postoperative antiemetics usage | 7 days
  The amount of rescue antiemetics given in the postoperative period, and until 7 days after surgery.
The inflammatory response expressed by C-reactive protein(CRP). | 2 days
  The inflammatory response is monitored by the blood-sample c-reactive protein(CRP) and analyzed to se the possible attenuation of the response because of dexamethasone.
Postoperative pain summarized in the first 7 days | 7 days
  Pain summarized over the first 7 days after surgery, assessed by a summation of the Visual Analog Scale(VAS)-scores in the first 7 days as noted in the pain diary filed in by the participants.
  Pain is monitored by the Visual Analog Scale(VAS) 0-100 mm, where 0 is no pain and 100 mm is the worst pain one can imagine. Moderate pain is considered a VAS >30 mm.

OTHER OUTCOMES:
Why still in hospital, an audit into the reasons the patient has not yet been discharged from the ward. | 7 days.
  An investigation into reason of why our patients remain in the hospital in the days after total Knee Arthroplasty in our Fast-Track center. This is investigated through a questionnaire previously used in a similar investigation in our center.
  The questionnaire is filled in by our project nurse. the questionnaire is a checkmark schedule with predetermined reasons to stay in hospital like low bloodpressure, sedation, dizzyness, lack of physiotherapy and medical and surgical complications.
  The outcome assesment will be descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Bang Foss, Dr.med., Study Director — Dept. of Anaesthesia, Hvidovre Hospital, Capital Region of Denmark.
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Capital Region of Denmark., Hvidovre
  - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen NI, Kehlet H, Gromov K, Troelsen A, Husted H, Varnum C, Kjaersgaard-Andersen P, Rasmussen LE, Pleckaitiene L, Foss NB. High-dose steroids in high pain responders undergoing total knee arthroplasty: a randomised double-blind trial. Br J Anaesth. 2022 Jan;128(1):150-158. doi: 10.1016/j.bja.2021.10.001. Epub 2021 Nov 5. PMID 34749994